CLINICAL TRIAL: NCT04541524
Title: Vienna Preserflo Microshunt Cohort Study
Brief Title: Vienna Preserflo Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Clemens Vass, Univ.Prof.Dr.med.univ., Medical University of Vienna
Other Study IDs: 1142_2020
Record Dates: First submitted 2020-07-17; First posted 2020-09-09 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Glaucoma; Glaucoma Surgery; Post-Op Complication; Efficacy, Self; Safety Issues
MeSH Terms: conditions — Glaucoma; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Device: Yes

INTERVENTIONS:
Device: Santen Preserflo Microshunt — The PMS is 8.5 mm long has an outer diameter of 350 μm and a lumen diameter of 70 μm. It has a fin sized 1.1 mm located 4.5 mm distally from the internal tip of the device and it consists of poly(styrene-b-isobutylene-b-styrene) SIBS. The device was implanted 1 year prior to the present study via an ab externo approach. At the beginning of the surgery, the conjunctiva was opened. In the first group of patients (group 1) we made a fornix based conjunctival opening, prepared a 1mm wide and long scleral pocket in 3mm distance from limbus and placed the PMS in the anterior chamber via a 25G needle track. In the second group (group 2) the conjunctival opening was 3.5 mm from the limbus, the scleral pocket was prepared at 3.5 mm distance from the limbus and a 27G needle was used. PMS guides aqueous humor from the anterior chamber to the subconjunctival space. The forming filtering bleb absorbs aqueous humor which leads to IOP reduction.

SUMMARY:
The Vienna Preserflo Microshunt Cohort Study is an observational study with a prospective postoperative examination in all glaucoma patients who had received a Preserflo Microshunt (PMS) as standalone procedure or in combination with cataract extraction in the time period between January and November 2019 at the Department of Ophthalmology, Medical University of Vienna. It is estimated that approximately 70 patients will be included of this cohort. The cohort will be invited for a prospective postoperative examination after 12 (±5) months of follow up. This examination shall comprise best corrected visual acuity, visual field test, intraocular pressure (IOP) measurement, slit lamp examination, fundus examination (optic disc and retina), gonioscopic assessment of PMS position, anterior segment optical coherence tomography (OCT) (shunt position, anterior chamber angle assessment, limbus shape analysis), corneal pachymetry, specular microscopy of corneal endothelial cells. Additionally, retrospective information concerning IOP, medication and visual fields of all patients will be collected from the Department of Ophthalmology as well as from the referring ophthalmologists where possible. Additionally, we will perform a comparison between two groups to compare differences in outcome measures.

DETAILED DESCRIPTION:
During the inclusion period two slightly different surgical approaches have been used. At the beginning of the surgery, the conjunctiva is opened and the Tenon capsule is getting dissected from the sclera. In the first group of patients (group 1) we made a fornix based conjunctival opening, prepared a 1mm wide and long scleral pocket in 3mm distance from limbus and placed the PMS in the anterior chamber via a 25G needle track. In the second group (group 2) the conjunctival opening was 3.5 mm from the limbus, the scleral pocket was prepared at 3.5 mm distance from the limbus and a 27G needle was used. The outcomes of these two groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Glaucoma patients who received a PMS in the time period between January and November 2019 at the Department of Ophthalmology, Medical University of Vienna, Austria, will be invited

Exclusion Criteria:

* Unwilling or unable to give informed consent.
* Pregnancy or lactation

Ages: 18 Years to 95 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Glaucoma patients who received a PMS as stndalone procedure or in combination with a cataract surgery in the time period between January and November 2019 at the Department of Ophthalmology, Medical University of Vienna, Austria, will be invited
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2020-06-05 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
IOP | one year
  IOP in mmHg
Full success | one year
  IOP below 21 and IOP reduction of at least 20% from baseline without medication
Qualified success | one year
  IOP below 21 and IOP reduction of at least 20% from baseline with or without medication
Complications | one year
  Number of complications per eye

SECONDARY OUTCOMES:
Re-intervention rate rate | one year
  Proportion of eyes requiring either needling revision of filtering bleb revision or any other glaucoma surgery
Medication rate | one year
  Number of patients who needed again eye pressure lowering medication
Average medication | one year
  Average number of different eye pressure lowering medication
OCT - shunt entry | one year
  Shunt position in chamber angle as determined by anterior segment OCT
OCT - shunt clearance | one year
  Shunt-cornea angle as determined by anterior segment OCT
OCT - shunt length | one year
  Shunt length in the anterior chamber as determined by anterior segment OCT
Corneal endothelial cell count | one year
  Corneal endothelial cell count in specular microscopy of corneal endothelium

CONTACTS AND LOCATIONS:
Locations (1):
- Insitute of Ophthalmology and Optometry, Medical University of Vienna, Vienna, Austria